CLINICAL TRIAL: NCT04920799
Title: Effect of Beet Juice Supplementation on Vascular and Inspiratory Muscle Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB202100040
Record Dates: First submitted 2021-05-27; First posted 2021-06-10 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate rich beetroot juice (Active Comparator)
  Interventions: Dietary Supplement: Nitrate rich beetroot juice
- Nitrate depleted beetroot juice (Placebo Comparator)
  Interventions: Dietary Supplement: Nitrate depleted beetroot juice

INTERVENTIONS:
Dietary Supplement: Nitrate rich beetroot juice — Participants will drink nitrate rich beetroot juice (2.4 floz ; Beet It Sport Nitrate 400 concentrated beetroot shot; James White Drink, ltd) twice daily for two weeks.
  Arms: Nitrate rich beetroot juice
Dietary Supplement: Nitrate depleted beetroot juice — Participants will drink nitrate depleted beetroot juice (2.4 floz ; Beet It placebo concentrated beetroot shot; James White Drink, ltd) twice daily for two weeks.
  Arms: Nitrate depleted beetroot juice

SUMMARY:
Older adults with coronary artery disease (CAD) have impaired vascular and inspiratory muscle function. The objective of this study is to examine the effect of beet juice supplementation on vascular and inspiratory muscle function in older adults with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Adults with coronary artery disease (CAD) based on an angiogram >50% stenosis in any major epicardial vessel or history of myocardial infarction or history of coronary revascularization.
* Considered to have stable CAD on optimal medical therapy
* 60 to 85 years of age
* Men and women (women must be postmenopausal either natural or surgical)
* Able to give consent

Exclusion Criteria:

* Ejection fraction <50%, unstable angina, recent myocardial infarction within 6 months
* Coronary revascularization, including percutaneous coronary intervention and coronary artery bypass graft or thoracic surgery within 6 months.
* Stroke, obstructive pulmonary disease, hepatitis B, C, HIV, seizures, or other relevant on-going or recurrent illness
* Individuals that have participated in respiratory training within the last 12 months or cardiac rehabilitation within the last 6 months
* Uncontrolled hypertension
* Use of tobacco products including smoking traditional or e-cigarettes
* Use of hormone replacement therapy in women or men (e.g., estrogen, progesterone or testosterone)
* Regular aerobic exercise training
* Unwilling to stop using mouthwash at least 1 week before the start of the study and during study participation
* Unwilling to remain weight stable during study participation

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in endothelial function | Baseline up to following 2 weeks of experimental condition
  Endothelial function will be determined using brachial artery flow-mediated dilation via high resolution duplex ultrasonography. Reactive hyperemia will be produced by inflating a forearm cuff to ~250 mmHg for 5 minutes followed by rapid deflation.
Change in inspiratory muscle function | Baseline up to following 2 weeks of experimental condition
  Inspiratory muscle function including strength, power and endurance will be assessed using the POWERbreathe KH2 device

SECONDARY OUTCOMES:
Change in microvascular function | Baseline up to following 2 weeks of experimental condition
  Microvascular function will be assessed using the forearm blood flow response to submaximal handgrip exercise. Brachial artery blood flow and diameter will be assessed using ultrasound.
Change in central arterial stiffness | Baseline up to following 2 weeks of experimental condition
  The SphygmoCor XCEL device will be used to measure carotid to femoral pulse wave velocity.
Change in central arterial hemodynamics | Baseline up to following 2 weeks of experimental condition
  The SphygmoCor XCEL device will be used to obtain central pulse wave analysis.
Change in functional capacity | Baseline up to following 2 weeks of experimental condition
  Using the Duke Activity Status Index we will assess participants' ability to perform daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Cardiovascular Physiology Laboratory, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No